CLINICAL TRIAL: NCT07145320
Title: The Impact of Oral Cryotherapy and Chewing Gum Interventions on Chemotherapy-induced Acute and Anticipatory Nausea, Vomiting, and Taste Alterations in Women Receiving Treatment for Breast Cancer: A Randomized Controlled Trial
Brief Title: The Impact of Oral Cryotherapy and Chewing Gum Interventions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Berna KURT, Assistant Professor, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KA-2020-05/615
Record Dates: First submitted 2025-08-08; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer; Nausea and Vomiting; Quality of Life; Chewing Gum
MeSH Terms: conditions — Breast Neoplasms; Nausea; Vomiting

STUDY DESIGN:
Intervention Model Description: This study employed a prospective, randomized controlled trial (RCT) design with three parallel arms to evaluate the efficacy of two non-pharmacologic interventions in managing chemotherapy-induced symptoms.
Who Masked: Investigator
Masking Description: All statistical analyses were carried out by an independent biostatistician blinded to group assignments to minimize bias and maintain analytical integrity.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Oral Cryotherapy Group (Group 1) (Experimental): Participants were educated about oral cryotherapy before their first chemotherapy cycle. Individually portioned ice bags (15 mL per cube) were prepared and provided free of charge for home use (6 bags per cycle). Patients were instructed to apply the ice intra-orally for 30 minutes at a time, 6-10 times daily, beginning at the start of Adriamycin infusion. A Cryotherapy Application Log Form was used to record date, start, and end times for each session.
  Interventions: Other: Oral Cryotherapy Group (Group 1)
- Chewing Gum Group (Group 2) (Experimental): Patients received standardized, tasteless, single-use chewing gum (6 boxes per cycle) and were instructed to chew a piece for 20-30 minutes before and during chemotherapy infusion. A new piece was provided midway through the session. Usage was recorded in a Chewing Gum Application Log Form, capturing date and timing details.
  Interventions: Other: Chewing Gum Group (Group 2)
- Control Group (Group 3) (No Intervention): Patients in the control group received routine clinical care and antiemetic treatment per protocol, with no additional interventions. Upon study completion, educational brochures and informational materials regarding oral cryotherapy and chewing gum interventions were provided to the control group to mitigate potential bias and ensure equitable access to relevant information.

INTERVENTIONS:
Other: Oral Cryotherapy Group (Group 1) — Participants were educated about oral cryotherapy before their first chemotherapy cycle. Individually portioned ice bags (15 mL per cube) were prepared and provided free of charge for home use (6 bags per cycle). Patients were instructed to apply the ice intra-orally for 30 minutes at a time, 6-10 times daily, beginning at the start of Adriamycin infusion. A Cryotherapy Application Log Form was used to record date, start, and end times for each session.
  Arms: Oral Cryotherapy Group (Group 1)
Other: Chewing Gum Group (Group 2) — Patients received standardized, tasteless, single-use chewing gum (6 boxes per cycle) and were instructed to chew a piece for 20-30 minutes before and during chemotherapy infusion. A new piece was provided midway through the session. Usage was recorded in a Chewing Gum Application Log Form, capturing date and timing details.
  Arms: Chewing Gum Group (Group 2)

SUMMARY:
Chemotherapy-induced nausea and vomiting (CINV) and taste alterations continue to be among the most common and most severe side effects that women receiving adjuvant chemotherapy for breast cancer suffer. Despite standard antiemetic treatments, a significant proportion of patients experience inadequate symptom management, necessitating investigation into complementary non-pharmacological interventions such as oral cryotherapy and chewing gum in women undergoing Adriamycin-Cyclophosphamide therapy. 135 female patients recently diagnosed with early-stage breast cancer participated in a single-center, three-arm randomized controlled trial. Random assignment was used to assign participants to the oral cryotherapy group (OCG), chewing gum group (CGG), or control group (CG). Interventions were used during the initial cycle of chemotherapy.

DETAILED DESCRIPTION:
Chemotherapy-induced nausea and vomiting (CINV) remains one of the most distressing and prevalent side effects of cancer treatment, affecting a substantial proportion of patients undergoing chemotherapy. Despite advances in antiemetic regimens, CINV continues to occur in many patients, significantly impairing their quality of life and clinical outcomes. The onset and severity of CINV are largely influenced by the emetogenic potential of chemotherapeutic agents, with drugs such as cyclophosphamide and doxorubicin frequently triggering acute symptoms within the first 1-5 days post-administration.

CINV is a multifactorial process involving both peripheral and central pathways. Cytotoxic agents stimulate the release of serotonin from enterochromaffin cells in the gastrointestinal tract, which subsequently activates 5-hydroxytryptamine 3 (5-HT₃) receptors in the chemoreceptor trigger zone (CTZ) of the central nervous system, leading to emesis. The CTZ, located in the area postrema of the medulla oblongata, is particularly vulnerable due to its lack of a complete blood-brain barrier, facilitating the access of circulating emetogenic substances. Beyond the immediate physical discomfort, poorly managed CINV contributes to complications including malnutrition, dehydration, electrolyte imbalances, metabolic disturbances, increased infection risk, and significant psychological distress. These complications often necessitate additional medical interventions and hospitalizations, increasing the financial and emotional burden on patients, caregivers, and healthcare systems. Despite routine pharmacologic interventions, many patients continue to experience CINV, which points to the importance of effective, accessible, and patient-centered non-pharmacologic approaches. Oral cryotherapy, localized cooling of the oral mucosa via ice application, has gained attention as a low-cost, well-tolerated method primarily used to prevent chemotherapy-induced oral mucositis. This method induces vasoconstriction of oral blood vessels during intravenous chemotherapy infusion, thereby limiting drug delivery to oral tissues. Although cryotherapy has been explored in other contexts, such as surgical nausea and gynecological care, its potential for CINV management remains underinvestigated. Another promising non-pharmacologic intervention is chewing gum, which stimulates salivary flow and may help mitigate the oral side effects of chemotherapy. Saliva has intrinsic protective and antimicrobial properties, and its production may be reduced by chemotherapy-induced cytotoxicity on salivary glands.

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 18 and 65 years,
* Scheduled to receive adjuvant chemotherapy for the first time,
* Receiving the AC protocol as their chemotherapy regimen,
* Receiving chemotherapy doses classified as moderately emetogenic (according to the International Society of Supportive Care in Cancer Guidelines),
* Not having received radiotherapy prior to adjuvant chemotherapy,
* Without chronic diseases (coronary artery disease, chronic kidney disease, or diabetes mellitus),
* Not having used any non-pharmacological method for nausea and vomiting,
* Diagnosed with breast cancer for the first time,
* Without metastasis,
* Without thrombocytopenia,
* At an early stage,
* Aware of their diagnosis,
* Open to communication and cooperation,
* Literate,
* Not receiving psychiatric and/or depression treatment,
* Not in the terminal stage,
* Willing and volunteering to participate in the study.

Exclusion Criteria:

* Illiterate,
* Over 65 years of age,
* Using anxiolytic or antidepressant medications,
* Having chronic diseases (gastrointestinal obstruction/disease, hepatitis, coronary artery disease, chronic kidney disease, or diabetes mellitus),
* Having metastasis,
* Having received radiotherapy prior to adjuvant chemotherapy,
* Not willing to participate in the study.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — 18-65
Enrollment: 135 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Chemotherapy-Induced Taste Alteration Scale (CITAS) | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Berna KURT, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Adnan Saygun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
will be shared upon request